CLINICAL TRIAL: NCT01330758
Title: A Phase I, Randomised, Open-label, Cross-over, Single-centre Study in Healthy Male and Non-fertile Female Volunteers to Determine the Relative Bioavailability of the Phase II Wet Granulation Tablet Formulation Compared to the Phase II/III Roller Compacted Tablet Formulation of AZD8931
Brief Title: A Study to Compare Two Different Tablet Formulations of AZD8931 in Healthy Males and Females
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Mary Stuart/Medical Science Director, AstraZeneca
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: D0102C00005
Record Dates: First submitted 2011-03-22; First posted 2011-04-07 (Estimated); Last update posted 2011-07-29 (Estimated); Status verified 2011-07

CONDITIONS: Healthy
Keywords: Phase I; Healthy male and non-fertile female volunteers; Bioavailability; AZD8931
MeSH Terms: interventions — AZD 8931

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 40 mg AZD8931 wet granulation tablet formulation (Active Comparator)
  Interventions: Drug: AZD8931
- 40 mg AZD8931 roller compacted tablet formulation (Experimental)
  Interventions: Drug: AZD8931

INTERVENTIONS:
Drug: AZD8931 — 40 mg AZD8931 wet granulation tablet formulation
  Arms: 40 mg AZD8931 wet granulation tablet formulation
Drug: AZD8931 — 40 mg AZD8931 roller compacted tablet formulation
  Arms: 40 mg AZD8931 roller compacted tablet formulation

SUMMARY:
A study to compare two different tablet formulations of AZD8931 in healthy males and females.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18 to 55 years
* Females must have a negative pregnancy test at screening and on admission to the unit, must not be lactating and must be of non-child bearing potential
* Body mass index between 19 and 30 kg/m2 and weight at least 50 kg and no more than 100 kg
* Male subjects must be willing to use barrier methods of contraception
* Be willing and able to comply with study procedures, restrictions and requirements

Exclusion Criteria:

* History of any clinically significant disease or disorder
* Any clinically significant abnormalities at screening
* Use of any prescribed or non-prescribed medication within 2 weeks
* Receipt of another NCE or participation in any other clinical trial within 3 months
* Subjects who have previously received AZD8931

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2011-04; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
To determine the relative bioavailability of 40 mg AZD8931 Phase II wet granulation tablet formulation in relation to the 40mg AZD8931 Phase II/III roller compacted tablet formulation. | Pharmacokinetic (PK) sampling will be performed day 1 to day 5 for each treatment period

SECONDARY OUTCOMES:
To further investigate the safety and tolerability variables (adverse events,vital signs, ECG, physical examination, safety labs). | From screening period through to 5 to 10 days after visit 3. An average time of 7 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Stuart, Study Director — AstraZeneca,1F64, Mereside, Alderley Park, Macclesfield, Cheshire,SK10 4TG UK; Dr Darren Wilbraham, DICP, MBBS, Principal Investigator — Quintiles Drug Research Unit at Guy's Hospital; Jason Clark, BSc, Study Director — Quintiles Drug Research Unit at Guy's Hospital
Locations (1):
- Research Site, London, United Kingdom